CLINICAL TRIAL: NCT00391352
Title: A Phase 4, fMRI Study of Treatment Recommendations Comparing Patients Taking IFN-β-1a 44 mcg Tiw SC (Rebif®) to Controls of Patients Recently Diagnosed With Relapsing Remitting Multiple Sclerosis Currently Naive to Disease-Modifying Therapy.
Brief Title: fMRI Study of Treatment Recommendations Comparing Recently Diagnosed Multiple Sclerosis (MS) Patients to Controls
Status: Completed | Type: Observational
Sponsor: Waukesha Memorial Hospital (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Michael McCrea, Waukesha Memorial Hospital
Other Study IDs: MSR12006
Record Dates: First submitted 2006-10-19; First posted 2006-10-23 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2008-05

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Disease Modifying Therapy
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MS: MS patient is matched to healthy volunteer
  Interventions: Drug: IFN-β-1a (Rebif®)
- Control

INTERVENTIONS:
Drug: IFN-β-1a (Rebif®) — 44 mcg Three times a week, subcutaneous injection
  Groups: MS

SUMMARY:
Impaired short term memory, attention and concentration lapses, and slower processing of information occur in up to 40-65% of patients with Multiple Sclerosis (MS). The quality of life of individuals with MS is impacted to the degree with which they experience these symptoms.

There are several medications approved by the United States Food and Drug Administration (FDA) to treat MS symptoms and to modify (slow) disease course. Traditional approaches to determining the effectiveness of medications used in treating MS rely on reports of the number of relapses an individual experiences, as well as standard clinical tests, such as the Kurtzke Expanded Disability Status Scale (EDSS).

This research study will look at whether the functional magnetic resonance imaging (fMRI) scan can be used as a tool for measuring changes in the brain associated with treatment in MS patients. Unlike a typical MRI which provides structural information about the brain, the fMRI provides information about brain activity during performance of cognitive or motor tasks.

DETAILED DESCRIPTION:
The development of the immunomodulatory, disease-modifying therapies (DMT) represents a major advance for the treatment of multiple sclerosis (MS). To date, immunomodulatory agents approved for the treatment of MS in the United States include two forms of recombinant interferon-beta (IFN-beta-1a [Avonex, Rebif] and IFN-beta-1b [Betaseron]) and synthetic glatiramer acetate [Copaxone]. These drugs have been shown to favorably alter the natural history of relapsing remitting MS by slowing the progression of disability, reducing relapse rate, and decreasing brain inflammation as measured by MRI. There is evidence that the treatment effects of both IFN-beta and glatiramer acetate are related to their properties in regulating various components of the immune system, in particular, the T cell functions (e.g. proliferation and migratory behavior) and cytokine production.

Though demonstrating clear efficacy on a number of short-term clinical measures, these agents are not cures and most patients with MS continue to experience disease activity in spite of treatment. Over the last ten years, clinicians have become comfortable initiating therapy with DMT. Now, attention is focused on monitoring the results of a chosen therapy and deciding whether or not a patient is responding optimally to treatment. At present, however, clinicians lack criteria for defining optimal response to DMT as well as evidence-based recommendations on how to improve treatment outcomes for individual patients.

Using a recently published model generated by an advisory board from the United States, as a framework, The Canadian Multiple Sclerosis Working Group (CMSWG) developed practical, evidence-based recommendations on how neurologists can assess the status of patients on DMT and decide when it may be necessary to modify treatment in order to optimize outcomes. The CMSWG's recommendations are based on monitoring relapses, neurological progression and MRI activity. These recommendations have yet to be implemented in a prospective, randomized, comparative Phase IV clinical trial.

Traditional measures do not provide critical information about the neural systems that underlie change in behavioral performance. The goal of developing a surrogate biological marker of drug efficacy is to be able to measure the extent to which a drug reaches its intended targeted neural system, and to understand and predict the impact of treatment on existing neuropathology. Ideally, relevant clinical outcome measures should be well correlated with the biomarker.

fMRI is a new tool for noninvasive imaging of human brain function. Without the use of contrast agents, fMRI detects regional MR signal increases that have been hypothesized to reflect decreases in deoxyhemoglobin due to local increases in blood flow/volume during task activation. fMRI has higher spatial and temporal resolution than other existing functional imaging techniques, making it ideal for the study of complex cognitive functions in patient populations.

ELIGIBILITY:
Inclusion Criteria MS Subjects:

* Written informed consent and HIPAA authorization.

  * Age between 18 and 65 years
  * Male and female subjects with clinically definite or laboratory-supported definite relapsing-remitting multiple sclerosis in accordance with the refined McDonald • Diagnosed with Relapsing-Remitting Multiple Sclerosis for ≤ 1 year
  * Naive to disease-modifying treatments
  * Expanded Disability Status Score (EDSS) of 0 to ≤ 5.5, inclusive
  * Willingness and ability to comply with the protocol for the duration of the study
  * If female, she must either:

    1. be post-menopausal or surgically sterilized; or
    2. use a hormonal contraceptive, intra uterine device, diaphragm with spermicide, or condom with spermicide, for the duration of the study; and
    3. be neither pregnant nor breast-feeding.
    4. confirmation that if the subject can still have children, that she is not pregnant must be established by a negative urine pregnancy test within 30 days of Study Day o.

Exclusion Criteria - MS Subjects:

* Pregnant or lactating women, or women of childbearing potential not using an acceptable method of contraception
* Progressive forms of MS (Primary progressive, Secondary progressive)
* Subjects who have been on DMTs or other previous treatment for MS
* Participation in any other studies involving investigational or marketed products, concomitantly or within 30 days prior to screening
* Treatment with oral or systemic corticosteroids or ACTH within 4 weeks of screening or ongoing chronic treatment with systemic corticosteroids.
* Have taken intravenous immunoglobulin or any other investigational drug or taken part in any experimental procedure in the 6 months prior to screening
* Psychiatric disorder either unstable or would preclude safe participation in the study
* Cognitive impairment which impairs ability to understand or comply with the protocol procedures
* Significant leucopenia (white blood cell count <0.5 times the lower limit of normal) as assessed during the course of routine standard of care
* Elevated liver function tests (ALT, AST, alkaline phosphatase or total bilirubin >2.5 times the upper limit of normal) as assessed during the course of routine standard of care
* Specific systemic diseases, (including insulin-dependent diabetes, Lyme disease, clinically significant cardiac disease, HIV, HTLV-1, and Hepatitis B or C), or other uncontrolled major medical conditions (depression, seizure disorder) that would interfere with the participant's safety, compliance or evaluation
* Unable and/or unlikely to follow the protocol for any reason
* Alcohol and/or any other drug abuse
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol.
* Abnormal baseline clinical findings considered by the investigator to be indicative of conditions that might affect study results
* Subjects whose high-resolution anatomic MR scans reveal the presence of a structural abnormality (other than MS)

Specific exclusion criteria are required for MRI scanning:

* Ferrous objects within the body
* Pregnancy
* Weight inappropriate for height
* Low visual acuity that cannot be corrected with glasses
* History of claustrophobia
* Standard protocol for monitoring based on FDA approved medication will be followed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ProHealth Care, Waukesha Memorial Hospital Neuroscience Center
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2008-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Primary: Examine the change in task-activated fMRI response as a function of disease modifying therapy assigned to MS as compared to controls | Week 24

SECONDARY OUTCOMES:
Neuropsychological and Neurological outcome measures. | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Michael McCrea, PhD, Principal Investigator — Waukesha Memorial Hospital; Stephen Rao, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Waukesha Memorial Hospital ProHealth Care, Waukesha, Wisconsin, United States